CLINICAL TRIAL: NCT02906813
Title: A Phase 1 Bioavailability and Food Effect Study to Compare Tablet Versus Solution Formulation and to Assess the Effect of Food on the Bioavailability of a Single TAK-935 Dose in Healthy Subjects
Brief Title: A Study to Determine the Bioavailability and Food Effect of a Single TAK-935 Dose in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-935-1005; U1111-1177-8044 (Registry Identifier: WHO)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-935 300 mg (Tablets Fed+Tablets Fasted+Solution Fasted) (Experimental): TAK-935 300 mg, tablets, orally, 30 minutes after a high-fat meal on Day 1 of Intervention Period 1, followed by a washout period of at least 3 days, further followed by TAK-935 300 mg, tablets, orally, under fasted state on Day 1 of Intervention Period 2, followed by a washout period of at least 3 days, further followed by TAK-935 300 mg, solution, orally, in fasted state on Day 1 of Intervention Period 3.
  Interventions: Drug: TAK-935 Tablets; Drug: TAK-935 Oral Solution
- TAK-935 300 mg (Tablets Fasted+Solution Fasted+Tablets Fed (Experimental): TAK-935 300 mg, tablets, orally under fasted state on Day 1 of Intervention Period 1, followed by a washout period of at least 3 days, further followed by TAK-935 300 mg, solution, orally, in fasted state on Day 1 of Intervention Period 2, followed by a washout period of at least 3 days, further followed by TAK-935 300 mg tablets, orally, 30 minutes after high-fat meal on Day 1 of Intervention Period 3.
  Interventions: Drug: TAK-935 Tablets; Drug: TAK-935 Oral Solution
- TAK-935 300 mg (Solution Fasted+Tablets Fed+Tablets Fasted) (Experimental): TAK-935 300 mg, solution, orally, in fasted state on Day 1 of Intervention Period 1, followed by washout period of at least 3 days, further followed by TAK-935 300 mg, tablets, orally, 30 minutes after a high-fat meal on Day 1 of Intervention Period 2, followed by washout period of at least 3 days, further followed by TAK-935 300 mg, tablets, orally, under fasted state on Day 1 of Intervention Period 3.
  Interventions: Drug: TAK-935 Tablets; Drug: TAK-935 Oral Solution

INTERVENTIONS:
Drug: TAK-935 Tablets — Tablets
Drug: TAK-935 Oral Solution — Oral solution

SUMMARY:
The purpose of this study is to assess the relative bioavailability (BA) of 300 milligram (mg) TAK-935 tablets compared to 300 mg of TAK-935 solution and to determine the effect of food on the BA of TAK-935 300 mg tablets in healthy adult participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-935. The study will look at the relative BA of TAK-935 300 mg tablets compared to a TAK-935 300 mg oral solution and will assess the effect of food on the BA of TAK-935 300 mg tablets in healthy adult participants.

The study will enroll approximately 9 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the 3 treatment sequences:

* TAK-935 (300 mg Tablets Fed + 300 mg Tablets Fasted + 300 mg Solution Fasted)
* TAK-935 (300 mg Tablets Fasted + 300 mg Solution Fasted + 300 mg Tablets Fed)
* TAK-935 (300 mg Solution Fasted + 300 mg Tablets Fed + 300 mg Tablets Fasted)

Administration of each dose will be separated by a washout period of at least 3 days. Participants will be asked to take single dose of TAK-935 tablet or oral solution on Day 1 of each Intervention Period.

This single center trial will be conducted in the United States. The overall time to participate in this study is 39 days. Participants will remain confined to the clinic from Day 1 of Intervention Period 1 to Day 3 of Intervention Period 3 and will be contacted by telephone 30 days after last dose of TAK-935 for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Weighs at least 45 kilogram (kg) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening and Day -2.

Exclusion Criteria:

1. Has received TAK-935 in a previous clinical study or as a therapeutic agent.
2. Has a history of any psychiatric disorder as diagnosed utilizing Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) criteria.
3. Has any lifetime history of drug abuse (defined as any illicit drug use) or any lifetime history of alcohol abuse prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or a single measure of spirits or 1 small glass of wine.
4. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
5. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody at Screening or a known history of human immunodeficiency virus infection.
6. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-In Day -1. Cotinine test is positive at Screening or Check-In (Day -1).
7. Has poor peripheral venous access.
8. Has donated or lost 450 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1 of Period 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 12 September 2016 to 09 November 2016.
Pre-assignment Details: Healthy participants were enrolled in 1 of the 3 treatment sequences that determined the order of the three treatments received: TAK-935 300 milligram (mg) tablets in fasted state, TAK-935 300 mg tablets in fed state and TAK-935 300 mg solution in fasted state.
Groups:
- TAK-935 300 mg: Tablets Fed + Tablets Fasted + Solution Fasted: TAK-935 3*100 mg, tablets, orally, 30 minutes after starting ingestion of a high-fat meal, once on Day 1 of Intervention Period 1, followed by a minimum 3-day washout period, further followed by TAK-935 3*100 mg, tablets, orally, after a 10-hour fast, once on Day 1 of Intervention Period 2, followed by a minimum 3-day washout period, further followed by TAK-935 300 mg, solution, orally, after a 10-hour fast, once on Day 1 of Intervention Period 3.
- TAK-935 300 mg: Tablets Fasted + Solution Fasted + Tablets Fed: TAK-935 3*100 mg, tablets, orally, after a 10-hour fast, once on Day 1 of Intervention Period 1, followed by a minimum 3-day washout period, further followed by TAK-935 300 mg, solution, orally, after a 10-hour fast, once on Day 1 of Intervention Period 2, followed by a minimum 3-day washout period, further followed by TAK-935 3*100 mg, tablets, orally, 30 minutes after starting ingestion of a high-fat meal, once on Day 1 of Intervention Period 3.
- TAK 935 300 mg: Solution Fasted + Tablets Fed + Tablets Fasted: TAK-935 300 mg, solution, orally, after a 10-hour fast, once on Day 1 of Intervention Period 1, followed by a minimum 3-day washout period, further followed by TAK-935 3*100 mg, tablets, orally, 30 minutes after starting ingestion of a high-fat meal, once on Day 1 of Intervention Period 2, followed by a minimum 3-day washout period, further followed by TAK-935 3*100 mg, tablets, orally, after a 10-hour fast, once on Day 1 of Intervention Period 3.
Period: Intervention Period 1 (3 Days)
Arm/Group | TAK-935 300 mg: Tablets Fed + Tablets Fasted + Solution Fasted | TAK-935 300 mg: Tablets Fasted + Solution Fasted + Tablets Fed | TAK 935 300 mg: Solution Fasted + Tablets Fed + Tablets Fasted
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period 1 (at Least 3 Days)
Arm/Group | TAK-935 300 mg: Tablets Fed + Tablets Fasted + Solution Fasted | TAK-935 300 mg: Tablets Fasted + Solution Fasted + Tablets Fed | TAK 935 300 mg: Solution Fasted + Tablets Fed + Tablets Fasted
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Intervention Period 2 (3 Days)
Arm/Group | TAK-935 300 mg: Tablets Fed + Tablets Fasted + Solution Fasted | TAK-935 300 mg: Tablets Fasted + Solution Fasted + Tablets Fed | TAK 935 300 mg: Solution Fasted + Tablets Fed + Tablets Fasted
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Washout Period 2 (at Least 3 Days)
Arm/Group | TAK-935 300 mg: Tablets Fed + Tablets Fasted + Solution Fasted | TAK-935 300 mg: Tablets Fasted + Solution Fasted + Tablets Fed | TAK 935 300 mg: Solution Fasted + Tablets Fed + Tablets Fasted
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0
Period: Intervention Period 3 (3 Days)
Arm/Group | TAK-935 300 mg: Tablets Fed + Tablets Fasted + Solution Fasted | TAK-935 300 mg: Tablets Fasted + Solution Fasted + Tablets Fed | TAK 935 300 mg: Solution Fasted + Tablets Fed + Tablets Fasted
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-935 300 mg: Tablets Fed + Tablets Fasted + Solution Fasted | TAK-935 300 mg: Tablets Fasted + Solution Fasted + Tablets Fed | TAK 935 300 mg: Solution Fasted + Tablets Fed + Tablets Fasted | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (7.77) | 37.0 (3.00) | 35.7 (13.58) | 36.7 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 0 | 5
  White | 0 | 1 | 2 | 3
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 9
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.0 (6.24) | 171.0 (2.00) | 170.3 (1.53) | 171.1 (3.44)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 83.17 (10.970) | 78.20 (1.311) | 71.50 (10.096) | 77.62 (9.039)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 28.01 (1.784) | 26.75 (0.889) | 24.62 (3.295) | 26.46 (2.430)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 2 | 2 | 3 | 7
  Ex-smoker | 1 | 1 | 0 | 2
No Alcohol Consumption [Count of Participants; unit: Participants] | 3 | 3 | 3 | 9
No Xanthine/Caffeine Consumption [Count of Participants; unit: Participants] | 3 | 3 | 3 | 9
Female Reproductive Status [Count of Participants; unit: Participants]
  Postmenopausal | 0 | 0 | 1 | 1
  Having childbearing potential | 1 | 0 | 0 | 1
  Not applicable | 2 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who were enrolled, received study drug and had at least 1 measurable plasma concentration for either TAK-935 or its metabolite (M-I).
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-935 300 mg Tablets Fed: TAK-935 3*100 mg, tablets, orally, 30 minutes after starting ingestion of a high-fat meal, once on Day 1 of either Intervention Period 1, 2 or 3.
- TAK-935 300 mg Tablets Fasted: TAK-935 3*100 mg, tablets, orally, after a 10-hour fast, once on Day 1 of either Intervention Period 1, 2 or 3.
- TAK-935 300 mg Solution Fasted: TAK-935 300 mg, solution, orally, after a 10-hour fast, once on Day 1 of either Intervention Period 1, 2 or 3.
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
Number analyzed (Participants) | 9 | 9 | 9
nanogram per milliliter (ng/mL) | 477.000 (298.0705) | 1150.889 (710.5940) | 1882.000 (1250.7022)
Statistical Analysis 1: Comparison: TAK-935 300 mg Tablets Fasted vs TAK-935 300 mg Solution Fasted; Analysis of variance (ANOVA) was performed on natural logarithms of TAK-935 Cmax with fixed factors of sequence, period and regimen, and random factor of participant nested within sequence. Pairwise comparisons was used to assess relative bioavailability (BA) of TAK-935 tablet to solution. Point estimate and 90 percent (%) confidence interval (CI) in original scale were obtained by exponentiation of differences in natural-log scale; Test type: Superiority or Other; p = 0.079, ANOVA; Least Square (LS) Mean Ratio = 0.631, 90% CI 2-sided [0.411 to 0.969]
Statistical Analysis 2: Comparison: TAK-935 300 mg Tablets Fed vs TAK-935 300 mg Tablets Fasted; ANOVA was performed on natural logarithms of TAK-935 Cmax with fixed factors of sequence, period, and regimen and random factor of participant nested within sequence. Pairwise comparisons was used to assess relative BA of TAK-935 administered after high-fat meal versus fasted. Point estimate and its 90% confidence interval in original scale were obtained by exponentiation of differences in natural-log scale; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean Ratio = 0.403, 90% CI 2-sided [0.262 to 0.618]

2. Primary Outcome: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK set included all participants who were enrolled, received study drug and had at least 1 measurable plasma concentration for either TAK-935 or its M-I.
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
Number analyzed (Participants) | 9 | 9 | 9
nanogram hours per milliliter (ng*hr/mL) | 1170.954 (386.1425) | 1328.482 (496.8168) | 1601.806 (711.7143)
Statistical Analysis 1: Comparison: TAK-935 300 mg Tablets Fasted vs TAK-935 300 mg Solution Fasted; ANOVA was performed on natural logarithms of TAK-935 AUCt with fixed factors of sequence, period, and regimen and random factor of participant nested within sequence. Pairwise comparisons was used to assess relative BA of TAK-935 tablet to solution. Point estimate and 90% CI in original scale were obtained by exponentiation of differences in natural-log scale; Test type: Superiority or Other; p = 0.146, ANOVA; LS Mean Ratio = 0.850, 90% CI 2-sided [0.706 to 1.024]
Statistical Analysis 2: Comparison: TAK-935 300 mg Tablets Fed vs TAK-935 300 mg Tablets Fasted; ANOVA was performed on natural logarithms of TAK-935 AUCt with factors of sequence, period, and regimen and random factor of participant nested within sequence. Pairwise comparisons was used to assess relative BA of TAK-935 administered after high-fat meal versus fasted. Point estimate and its 90% CI in original scale were obtained by exponentiation of differences in natural-log scale; Test type: Superiority or Other; p = 0.281, ANOVA; LS Mean Ratio = 0.889, 90% CI 2-sided [0.738 to 1.070]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-935
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK analysis set where data on Day 1 was available. The PK set included all participants who were enrolled, received study drug and had at least 1 measurable plasma concentration for either TAK-935 or its M-I.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
Number analyzed (Participants) | 9 | 8 | 8
ng*hr/mL | 1182.641 (385.6485) | 1369.963 (523.2334) | 1564.307 (743.3798)
Statistical Analysis 1: Comparison: TAK-935 300 mg Tablets Fasted vs TAK-935 300 mg Solution Fasted; ANOVA was performed on natural logarithms of TAK-935 AUC∞ with fixed factors of sequence, period, and regimen and random factor of participant nested within sequence. Pairwise comparisons was used to assess relative BA of TAK-935 tablet to solution. Point estimate and 90% CI in original scale were obtained by exponentiation of differences in natural-log scale; Test type: Superiority or Other; p = 0.191, ANOVA; LS Mean Ratio = 0.842, 90% CI 2-sided [0.676 to 1.050]
Statistical Analysis 2: Comparison: TAK-935 300 mg Tablets Fed vs TAK-935 300 mg Tablets Fasted; ANOVA was performed on natural logarithms of TAK-935 AUC∞ with factors of sequence, period, and regimen and random factor of participant nested within sequence. Pairwise comparisons was used to assess relative BA of TAK-935 administered after high-fat meal versus fasted. Point estimate and its 90% CI in original scale were obtained by exponentiation of differences in natural-log scale; Test type: Superiority or Other; p = 0.355, ANOVA; LS Mean Ratio = 0.894, 90% CI [0.726 to 1.100]

4. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to 30 days after last dose of study drug (Day 39)
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 0 | 22.2 | 0

5. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Time Frame: Baseline up to Day 11
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose.
Time Frame: Baseline up to Day 11
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 22.2 | 0 | 33.3

7. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Post Dose
Time Frame: Baseline up to Day 11
Population: The safety analysis set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 33.3 | 33.3 | 55.6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days (Day 39) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-935 300 mg Tablets Fed | TAK-935 300 mg Tablets Fasted | TAK-935 300 mg Solution Fasted
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 2/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-935 300 mg Tablets Fed (N=9) | TAK-935 300 mg Tablets Fasted (N=9) | TAK-935 300 mg Solution Fasted (N=9)
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.